CLINICAL TRIAL: NCT07263711
Title: A Prospective Real-World Study of Pathology Artificial Intelligence for Predicting Molecular Alterations in Gliomas
Brief Title: Prospective Real-World Study of Pathology AI for Glioma Molecular Prediction
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-508
Record Dates: First submitted 2025-11-13; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical study is to learn if an artificial intelligence (AI) model can accurately predict important molecular changes in gliomas, a type of brain tumor, using digital pathology images.

The main questions this study aims to answer are:

How accurate is the AI model in predicting key molecular alterations compared with standard molecular testing? Can the AI model shorten the time needed for diagnosis and reduce the need for expensive molecular tests?

Researchers will collect whole slide images from multiple hospitals and use the AI model to predict molecular results. The predictions will be compared with the actual test results from standard laboratory methods.

Participants will:

Allow the use of their pathology images and molecular test results for research.

Have no additional treatments or procedures beyond standard medical care.

This study will help determine whether AI-assisted tools can provide faster and lower-cost molecular diagnosis for glioma, improving patient care and supporting equal access to precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or legally authorized representative) has voluntarily signed the informed consent form.
* Age ≥ 18 years at the time of enrollment.
* Histologically suspected diffuse glioma based on biopsy or surgical resection.
* Availability of complete clinical information and usable digital pathology slides with hematoxylin and eosin (H&E) staining.
* Postoperative molecular pathology results available for comparison.

Exclusion Criteria:

* Poor-quality pathology samples (e.g., insufficient tissue, large folding or contamination of slides, or substandard digital scanning quality).
* Determined by the investigator to be unsuitable for participation in the study for any reason.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult participants (aged 18 years or older) who have been diagnosed with or are suspected to have diffuse glioma based on biopsy or surgical resection. Participants must have available hematoxylin and eosin (H&E)-stained digital pathology slides and complete clinical and molecular testing data.
  All participants will be patients who have received standard medical care for glioma. No additional treatments or interventions will be performed as part of this study. Pathology images and molecular testing results will be collected prospectively from multiple clinical centers to evaluate the diagnostic performance of the AI-based pathology model.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI model in predicting key molecular alterations in glioma | Within 1 week after whole slide images (WSIs) are obtained
  The primary outcome is the diagnostic performance of the AI-based pathology model in predicting key molecular alterations in glioma. Accuracy, sensitivity, specificity, and area under the receiver operating characteristic curve (AUC) will be calculated by comparing AI predictions with reference results from standard molecular pathology testing.

CONTACTS AND LOCATIONS:
Overall Officials: LI LIANG, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China